CLINICAL TRIAL: NCT00152841
Title: Effect of Iron and Antioxidant Vitamins on Disease Activity and Oxidative Stress in Inflammatory Bowel Disease (IBD)
Brief Title: Effect of Iron and Vitamin E Supplementation on Disease Activity in Patients With Either Crohn's Disease or Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patients
Sponsor: University Health Network, Toronto (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Dr. Johane Allard, Toronto General Hospital- UHN
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 02-0289-E
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Mild or Moderate Anaemia
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Lymphoma, Follicular | interventions — Iron-Dextran Complex; Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Iron supplement 300-600 mg/day
Drug: Vitamin E 800IU

SUMMARY:
Hypothesis:In patients with ulcerative colitis and Crohn's disease diagnosed with mild or moderate anaemia:

1. iron supplementation will increase disease activity and oxidative stress
2. the addition of antioxidant vitamin will reduce this detrimental effect

DETAILED DESCRIPTION:
To maintain site/extent of disease and medication consistent among groups, the design is a double blind crossover placebo-controlled trial.

1. If mild anaemia, patients are randomized to 300 mg of ferrous fumarate or placebo for 4 weeks followed by 2 weeks of washout period after which patients will crossover the opposite treatments for another 4 weeks.
2. If moderate anaemia, patients will receive 600 mg of ferrous fumarate for 10 weeks. They are randomized to either vitamin E (800 IU) or placebo for 4 weeks followed by 2 weeks of washout period after which patients will crossover the opposite treatments for another 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* diagnosed with inflammatory Bowel Disease (ulcerative colitis and Crohn's disease)
* with mild or moderate anaemia

Exclusion Criteria:

* not diagnosed with bowel obstruction
* not diagnosed with short bowel syndrome
* not taking iron supplement or antioxidant vitamins and minerals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2002-06; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
calprotectin in stools at baseline, week 4, week 6, week 10

SECONDARY OUTCOMES:
disease activity index
oxidative stress (plasma lipid peroxides, antioxidant potency, vitamin C, vitamin E, superoxide dismutase)
blood measurement of CBD
iron status

CONTACTS AND LOCATIONS:
Overall Officials: Allard Johane, MD, FRCPC, Principal Investigator — University Health Network - Toronto General Hospital
Locations (1):
- University Health Network - Toronto General Hospital, Toronto, Ontario, Canada